CLINICAL TRIAL: NCT00421655
Title: A Phase III Trial Assessing the Efficacy and Safety of Grazax in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: A Trial of Grazax in Subjects With Hayfever
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Kim Simonsen, MD, Senior Director, ALK-Abello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-14
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Grazax

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Grazax
- 2 (Placebo Comparator)
  Interventions: Drug: Grazax

INTERVENTIONS:
Drug: Grazax — Tablets 75,000 SQT and matching placebo. One tablet daily.

SUMMARY:
The trial is performed to evaluate the efficacy and safety of specific immunotherapy with Grazax for treatment of grass pollen induced allergy.

ELIGIBILITY:
Inclusion Criteria:

* History of grass pollen allergy
* Positive skin prick test to grass
* Positive specific IgE to grass

Exclusion Criteria

* FEV1 <70% of predicted value

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Recording of allergy symptoms | Grass pollen season 2007

CONTACTS AND LOCATIONS:
Overall Officials: Kim Simonsen, MD, Study Director — ALK-Abelló A/S
Locations (1):
- CompleWare Corporation, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Murphy K, Gawchik S, Bernstein D, Andersen J, Pedersen MR. A phase 3 trial assessing the efficacy and safety of grass allergy immunotherapy tablet in subjects with grass pollen-induced allergic rhinitis with or without conjunctivitis, with or without asthma. J Negat Results Biomed. 2013 Jun 1;12:10. doi: 10.1186/1477-5751-12-10. PMID 23725348